CLINICAL TRIAL: NCT00371059
Title: Pragmatic Randomized Control Trial of Memantine For Agitation In Dementia
Brief Title: Memantine for Agitation in Dementia
Acronym: MAGD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: East Kent Hospitals University NHS Foundation Trust (Other Government)
Collaborators: University of Oxford (Other); Institute of Psychiatry, London (Other); University of London (Other); University College, London (Other); Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005-005087-93; ISRCTN 24953404
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: DEMENTIA
Keywords: Agitation; Dementia; Alzheimer's
MeSH Terms: conditions — Dementia; Psychomotor Agitation | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Memantine — Memantine 10mg BD
Drug: Placebo — Placebo 10 mgs BD

SUMMARY:
We plan to evaluate the use of memantine in Alzheimer's disease to control agitation in the acute situation i.e under 12 weeks

DETAILED DESCRIPTION:
Agitation is a cause of morbidity and mortality in Alzheimer's due to distress and use of medication with side effects. Memantine has beed shown to be associated with less agitation and a recent study by forrest pharmaceuticals failed to recruit. We will perform a 12 week rct in 164 patients to test this hypothesis in a locality with no competing studies and in a clinical setting where the drug is not often used. We will compare with placebo and also use a rescue protocol derived from international best practice.

ELIGIBILITY:
Inclusion Criteria:

1. Residential/Inpatients at recruitment to the study with a history of at least 2 weeks behavioural disturbance.
2. Alzheimer's Disease only as per McKhann Criteria + Hachinski Score<=4.
3. Moderately severe to severe Alzheimer's Disease (baseline MMSE </=19).
4. Clinically significant agitation that requires treatment.
5. Severity of agitation defined by Cohen Mansfield agitation inventory (CMAI) > /=45.
6. Age >/= 55.

Exclusion Criteria:

1. Memantine usage in the 4 weeks prior to the start of the study.
2. On Cholinesterase inhibitor for less than 3 months and not on a stable dose.
3. Anti-psychotic, anti-epileptic, antidepressant, benzodiazepine, lithium or hypnotic dosage alteration in the 2 weeks prior to the start of the study.
4. Antiparkinsonian medication.
5. Hypersensitivity to memantine or any of the excipients in the formulation.
6. Severe renal impairment.
7. Epilepsy, history of convulsions or seizure, or receiving any anti-epileptic treatment.
8. Concomitant usage of N-methyl-D-aspartate (NMDA) antagonists such as amantadine, ketamine or dextromethorphan.
9. Recent myocardial infarction, uncompensated congestive heart failure and uncontrolled hypertension.
10. Severe, unstable or poorly controlled medical illness.
11. Any disability that may interfere with the patient completing the study procedure.
12. Active malignancy.
13. Delirium, pain or any medical illness as a clear cause of agitation.
14. Any important drug interactions: Prohibited during study and in the 14 days preceding enrollment/inclusion are: Analgesic dextromethorphan, Dopaminergics- amantadine, Warfarin due to theoretical INR prolongation.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Cohen-Mansfield | 2 weeks

SECONDARY OUTCOMES:
Neuropsychiatric Inventory 6+12 weeks | 2 weeks
Clinical Global Impression 6+ 12 weeks | 2 weeks
Severe Impairment Battery 6+12 weeks | 2 weeks
Quality of Life 6+12 weeks | 2 weeks
Co-meds | 2 weeks
Incidents of agitation | 2 weeks
Use of rescue protocol | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: CHRIS FOX, MBBSBscMSC, Principal Investigator — KENT AND MEDWAY NHS AND SOCIAL CARE PARTNERSHIP TRUST
Locations (2):
- United Kingdom (2):
  - Oxleas Nhs Foundation Trust, Dartford, KENT
  - Kent and Medway NHS and Social Care Partnership Trust, Folkestone, Kent

REFERENCES:
- [Derived] Fox C, Crugel M, Maidment I, Auestad BH, Coulton S, Treloar A, Ballard C, Boustani M, Katona C, Livingston G. Efficacy of memantine for agitation in Alzheimer's dementia: a randomised double-blind placebo controlled trial. PLoS One. 2012;7(5):e35185. doi: 10.1371/journal.pone.0035185. Epub 2012 May 2. PMID 22567095